CLINICAL TRIAL: NCT04567264
Title: Prospective Single Centre Trial of Percutaneous Tibial Nerve Stimulation With the Implantable StimRouter Neuromodulation System for the Treatment of Refractory Lower Urinary Tract Symptoms in Patients With Multiple Sclerosis
Brief Title: Wireless, Implantable Tibial Nerve Stimulator System for the Treatment of Refractory Lower Urinary Tract Symptoms in Patients With Multiple Sclerosis
Acronym: Stimrouter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiara Zecca (Other)
Collaborators: ABREOC (Unknown)
Responsible Party: Sponsor-Investigator, Chiara Zecca, Principal Investigator, Deputy Head of Multiple Sclerosis Center, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOC.NEUUR.2002
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: overactive bladder; posterior tibial nerve stimulation; lower urinary tract symptoms
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, single center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- With stimulation (Experimental): Implantation of device electrodes subcutaneous in lower tibia area; stimulation of posterior tibial nerves.
  Interventions: Device: StimRouter®, Self-activated and self-controlled neuromodulation device (Bioness Inc, CE0086).

INTERVENTIONS:
Device: StimRouter®, Self-activated and self-controlled neuromodulation device (Bioness Inc, CE0086). — Regimen 1 (weeks 0-12): one stimulation every 2 days, for a duration of 30 minutes each.
  Regimen 2 (weeks 12-24): Three stimulation treatments per week, for a duration of 30 minutes each.

SUMMARY:
Prevalence of lower urinary tract symptoms (LUTS) in patients with multiple sclerosis (MS) increases with disease duration. Current management of urinary clinical symptoms in MS is mainly conservative. Its long-term outcome is often poor because of the progressive disease course and the treatment related side effects. Alternative therapeutic options are botulinum toxin injections, electrical stimulation of dorsal penile/clitoral nerve, and sacral nerve modulation. Posterior tibial nerve stimulation (PTNS) is a second minimally invasive method of electrical stimulation. Multiple benefits may derive from the development and validation of a dedicated protocol of a new self-activated neuromodulation therapy, which may improve therapy compliance/effectiveness, quality of life and social life in MS patients with refractory LUTS. Furthermore, it may contribute to reduce outpatient visits, health costs and work absenteeism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 - 80;
2. Diagnosis of multiple sclerosis according to McDonald [20];
3. Clinical stability over the past 6 months (no relapses and no disability progression, defined as worsening of ≥1 point in the EDSS score if reference EDSS is ≤5.5, and ≥0.5 points if reference EDSS is>5.5);
4. One or more of: urinary frequency greater than 8 times/24 hours, urinary urge incontinence at least 2 episodes in 24 hours on 3-day voiding diary;
5. Urodynamic diagnosis of detrusor over-activity (DOA)and / or detrusor-sphincter dyssynergia (DSD);
6. Previous failure of conservative treatments (challenge over ≥6 months) i.e. lifestyle modification-fluid consumption, behavioral modification, and pharmacological therapy and stable OAB medications for at least 30 days;
7. No pharmacological treatment of overactive bladder (antimuscarinics and beta-3 agonists) for 2 weeks prior to screening;
8. Positive response to ongoing PTNS treatment defined as ≥50% reduction in urinary frequency, and/or ≥50% fewer incontinence episodes, or a return to normal voiding frequency (<8 voids/day), based on retrospective diary review (treatment compliant and non-compliant patients) or PTNS treatment naïve able to sense tibial nerve stimulation (to be tested with TENS exam).
9. Competent sphincter mechanism and normally functioning upper urinary tract;
10. Leg circumference in the range of 20-30 cm at implantation site;
11. No contraindications for surgical intervention (e.g. being immunocompetent, no anticoagulant treatment, no current infection);
12. For female patients: using effective contraceptive methods;
13. Ability to comply with study requirements;
14. Having provided written informed consent.

Exclusion Criteria:

1. Previous participation in another study with any investigational drug or device within the past 90 days;
2. Any metal implant in the area of StimRouter lead implantation site;
3. Anatomical defects that preclude use of the device;
4. Treatment with botulinum toxin injections, urinary incontinence surgery or implantation of artificial graft material, spinal or genitourinary surgery, abdominoperineal resection of the rectum or radical hysterectomy (female)/ prostatectomy (male) within the last 6 months;
5. Previous treatment with sacral neuromodulation;
6. Diagnosis of pelvic pain disorders, stress incontinence, current urinary tract infection, urinary stone and/or urinary tract malignancy; cystocele, enterocele or rectocele of grade 3 or 4;
7. Critical limb ischemia;
8. Previous or current pelvic radiotherapy and/or chemotherapy;
9. Severe uncontrolled diabetes;
10. Being prone to excessive bleeding;
11. Having a pacemaker or implantable defibrillator or other neural stimulation systems;
12. Exposure to diathermy or electrocautery;
13. Clinically significant peripheral neuropathy;
14. Neutropenic or immune compromised;
15. Pelvic radio- and/or chemotherapy;
16. Morbid obesity (BMI >40);
17. Pregnant or lactating women, or women planning a pregnancy during the study, <9 months post-partum;
18. Male: alpha-blocker for benign prostatic hyperplasia;
19. Allergy to local anesthetic or adhesive;
20. Life expectancy <1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in bladder volume | 6 months
  filling volume at the time of the first uninhibited detrusor contraction during cystometry

SECONDARY OUTCOMES:
Cystometric capacity (mL) | 6 months
  Video-urodynamic parameter
Compliance (ml/cmH20) | 6 months
  Video-urodynamic parameter
Maximum detrusor pressure (cmH20) during storage phase | 6 months
  Video-urodynamic parameter
Maximum detrusor pressure (cmH20) during voiding phase | 6 months
  Video-urodynamic parameter
Voided volume (mL) | 6 months
  Video-urodynamic parameter
Maximum flow rate (mL/s) | 6 months
  Video-urodynamic parameter
Post void residual | 6 months
  Video-urodynamic parameter
Pelvic floor electromyographic activity (normal/detrusor sphincter dyssynergia/non-relaxing pelvic floor) | 6 months
  Video-urodynamic parameter
Number of voids/day | 3, 4.5, 6 months
  3-day voiding diary
Volume voided/void | 3, 4.5, 6 months
  3-day voiding diary
Number of leaks per day | 3, 4.5, 6 months
  3-day voiding diary
Degree of urgency prior to void | 3, 4.5, 6 months
  3-day voiding diary
Number of CISC through the day | 3, 4.5, 6 months
  3-day voiding diary
Residual urine volume | 3, 4.5, 6 months
  3-day voiding diary
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 3, 4.5, 6 months
  54 items, two summary scores: physical health and mental health, range 0-100, a higher score indicates a better quality of life
Over active bladder questionnaire (OAB) | 3, 4.5, 6 months
  Symptom severity of OAB range 6-36, higher score values indicate greater symptom severity or bother, lower scores indicate minimal symptom severity.
  Health related quality of life (HRQL) subscales (coping, sleep, and social), range 13-78, Higher scores indicate better HRQL.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Lugano, Neurocenter of Southern Switzerland, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No